CLINICAL TRIAL: NCT03440385
Title: Induction Study #2 - A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Oral Ozanimod as Induction Therapy for Moderately to Severely Active Crohn's Disease
Brief Title: Induction Study #2 of Oral Ozanimod as Induction Therapy for Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-3202; U1111-1203-7949 (Registry Identifier: WHO); 2017-004293-33 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Crohn Disease; Oral; Ozanimod; Moderately active; Severely active; RPC01; RPC01-3202
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Administration of oral Ozanimod (Experimental)
  Interventions: Drug: Ozanimod
- Administration of Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Arms: Administration of oral Ozanimod
Other: Placebo — Specified dose on specified days
  Arms: Administration of Placebo

SUMMARY:
This is a study to explore the effect of oral ozanimod as an induction treatment for participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Crohn's disease for ≥ 3 months on endoscopy and on histological exam
* Inadequate response or loss of response to corticosteroids, immunomodulators, and/or biologic therapy
* Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450
* Average daily stool frequency ≥ 4 points and/or an abdominal pain of ≥ 2 points
* Simple Endoscopic Score for Crohn's Disease (SES-CD) score of ≥ 6 (or SES-CD ≥ 4 in participants with isolated ileal disease)

Exclusion Criteria:

* Diagnosis of ulcerative colitis, indeterminate colitis, radiation colitis, or ischemic colitis, or has strictures with prestenotic dilatation requiring procedural intervention
* Extensive small bowel resection (>100cm) or known diagnosis of short bowel syndrome, or requires total parenteral nutrition
* Current stoma, ileal-anal pouch anastomosis, or fistula

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (368):
- United States (81):
  - Local Institution - 202, Scottsdale, Arizona
  - Ucsd Medical Center, La Jolla, California
  - Local Institution - 010, Lancaster, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Matrix Clinical Research Inc, Los Angeles, California
  - Facey Medical Foundation (Parent), Mission Hills, California
  - Local Institution - 093, Pasadena, California
  - Sutter Medical Group, Roseville, California
  - Local Institution - 280, Sacramento, California
  - Local Institution - 281, San Francisco, California
  - Local Institution - 124, West Covina, California
  - Local Institution - 065, Colorado Springs, Colorado
  - Local Institution - 182, Bristol, Connecticut
  - Local Institution - 166, Clearwater, Florida
  - Local Institution - 084, Clermont, Florida
  - American Research Institute Inc, Cutler Bay, Florida
  - Local Institution - 112, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - SIH Research, Kissimmee, Florida
  - Local Institution - 067, Lighthouse PT, Florida
  - Center For Advanced Gastroenterology, Maitland, Florida
  - LMG Research, Miami, Florida
  - Local Institution - 175, Miami, Florida
  - Local Institution - 081, Miami, Florida
  - Local Institution - 044, Miami Springs, Florida
  - Local Institution - 192, New Port Richey, Florida
  - Local Institution - 200, Orlando, Florida
  - Local Institution - 002, Palmetto Bay, Florida
  - Theia Clinical Research, LLC, Pinellas Park, Florida
  - Precision Clinical Research, LLC., Sunrise, Florida
  - Local Institution - 183, Tampa, Florida
  - Apex Clinical Research, Tampa, Florida
  - Local Institution - 107, Tampa, Florida
  - Local Institution - 037, Atlanta, Georgia
  - Local Institution - 220, Atlanta, Georgia
  - Local Institution - 143, Decatur, Georgia
  - Local Institution - 115, Idaho Falls, Idaho
  - Local Institution - 022, Chicago, Illinois
  - Local Institution - 092, Evansville, Indiana
  - Local Institution - 033, Indianapolis, Indiana
  - Local Institution - 070, Topeka, Kansas
  - Local Institution - 020, Baton Rouge, Louisiana
  - Clinical Trials of SW Louisiana LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Local Institution - 024, Worcester, Massachusetts
  - Local Institution - 167, Kalamazoo, Michigan
  - Local Institution - 005, Novi, Michigan
  - Local Institution - 095, Minneapolis, Minnesota
  - Local Institution - 045, Rochester, Minnesota
  - Local Institution - 198, Kansas City, Missouri
  - Internal Medicine Specialists, Las Vegas, Nevada
  - Local Institution - 040, Lebanon, New Hampshire
  - Local Institution - 054, Hartsdale, New York
  - Weill Cornell Medical College, New York, New York
  - Concorde Medical Group, New York, New York
  - TrialSpark, New York, New York
  - Local Institution - 060, North Massapequa, New York
  - Local Institution - 156, Charlotte, North Carolina
  - Local Institution - 052, Winston-Salem, North Carolina
  - Local Institution - 170, Dayton, Ohio
  - Local Institution - 049, Hilliard, Ohio
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Local Institution - 087, Norman, Oklahoma
  - Local Institution - 294, Oklahoma City, Oklahoma
  - Local Institution - 185, Tulsa, Oklahoma
  - Local Institution - 217, Tulsa, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 034, Fort Sam Houston, Texas
  - Local Institution - 079, Houston, Texas
  - Local Institution - 196, Houston, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Accurate Clinical Research Inc, Pasadena, Texas
  - Local Institution - 071, Richardson, Texas
  - Local Institution - 178, San Antonio, Texas
  - Local Institution - 181, Temple, Texas
  - Local Institution - 292, Riverton, Utah
  - Local Institution - 030, Lynchburg, Virginia
  - The Gastroenterology Group, Reston, Virginia
  - Local Institution - 072, Richmond, Virginia
  - Local Institution - 172, Roanoke, Virginia
  - Local Institution - 089, La Crosse, Wisconsin
- Australia (13):
  - Local Institution - 309, Liverpool, New South Wales
  - Local Institution - 318, New Lambton Heights, New South Wales
  - Local Institution - 328, Herston, Queensland
  - Local Institution - 313, Maroorchydore, Queensland
  - Local Institution - 321, North Mackay, Queensland
  - Local Institution - 312, South Brisbane, Queensland
  - Local Institution - 307, Bedford Park, South Australia
  - Local Institution - 326, Elizabeth Vale, South Australia
  - Local Institution - 317, Clayton, Victoria
  - Local Institution - 305, Fitzroy, Victoria
  - Local Institution - 329, Geelong, Victoria
  - Local Institution - 327, Melbourne, Victoria
  - Local Institution - 315, Subiaco, Western Australia
- Austria (4):
  - Local Institution - 726, Innsbruck
  - Local Institution - 727, Sankt Pölten
  - Local Institution - 336, Vienna
  - Local Institution - 725, Vienna
- Bulgaria (6):
  - Local Institution - 753, Rousse
  - Local Institution - 750, Sofia
  - Local Institution - 755, Sofia
  - Local Institution - 756, Sofia
  - Local Institution - 752, Sofia
  - Local Institution - 554, Sofia
- Canada (9):
  - Local Institution - 269, Edmonton, Alberta
  - Local Institution - 262, New Westminster, British Columbia
  - Local Institution - 267, Vancouver, British Columbia
  - Local Institution - 256, Brandon, Manitoba
  - Local Institution - 266, Greater Sudbury, Ontario
  - Local Institution - 264, Toronto, Ontario
  - Local Institution - 257, Toronto, Ontario
  - Local Institution - 254, Montreal, Quebec
  - Local Institution - 270, Ottawa, Quebec
- China (35):
  - Local Institution - 423, Changzhou, Jiangsu
  - Local Institution - 369, Shanghai, Shanghai Municipality
  - Local Institution - 482, Beijing
  - Local Institution - 467, Beijing
  - Local Institution - 379, Bengbu
  - Local Institution - 485, Changchun
  - Local Institution - 376, Changchun
  - Local Institution - 421, Changsha
  - Local Institution - 378, Changsha
  - Local Institution - 414, Changzhou
  - Local Institution - 419, Chengdu
  - Local Institution - 422, Fuzhou
  - Local Institution - 478, Guangzhou
  - Local Institution - 472, Guangzhou
  - Local Institution - 486, Guangzhou
  - Local Institution - 470, Hangzhou, Zhejiang
  - Local Institution - 491, Hefei
  - Local Institution - 374, Kunming
  - Local Institution - 383, Luzhou
  - Local Institution - 488, Nanchang
  - Local Institution - 418, Nanjing
  - Local Institution - 375, Nanjing
  - Local Institution - 487, Nanjing
  - Local Institution - 473, Shanghai
  - Local Institution - 380, Shanghai
  - Local Institution - 377, Shanghai
  - Local Institution - 458, Taichung City
  - Local Institution - 373, Tianjin
  - Local Institution - 475, Wuhan
  - Local Institution - 474, Wuhan
  - Local Institution - 483, Wuhan
  - Local Institution - 381, Wuxi
  - Local Institution - 415, Xi'an
  - Local Institution - 420, Xi'an
  - Local Institution - 370, Zhengzhou
- Colombia (5):
  - Local Institution - 397, Armenia
  - Local Institution - 398, Barranquilla
  - Local Institution - 395, Bogotá
  - Local Institution - 396, Cali
  - Local Institution - 394, Medellín
- Finland (2):
  - Local Institution - 613, Helsinki
  - Local Institution - 614, Turku
- France (8):
  - Local Institution - 647, Neuilly-sur-Seine, Cedex
  - Local Institution - 639, Béziers
  - Local Institution - 635, Blois
  - Local Institution - 634, Caen
  - Local Institution - 644, Colombes
  - Local Institution - 632, Nantes
  - Local Institution - 630, Pierre-Bénite
  - Local Institution - 631, Saint-Priest-en-Jarez
- Georgia (15):
  - Local Institution - 786, Batumi
  - Local Institution - 779, Kutaisi
  - Local Institution - 454, Tbilisi
  - Local Institution - 778, Tbilisi
  - Local Institution - 782, Tbilisi
  - Local Institution - 552, Tbilisi
  - Local Institution - 793, Tbilisi
  - Local Institution - 740, Tbilisi
  - Local Institution - 783, Tbilisi
  - Local Institution - 784, Tbilisi
  - Local Institution - 785, Tbilisi
  - Local Institution - 335, Tbilisi
  - Local Institution - 455, Tbilisi
  - Local Institution - 781, Tbilisi
  - Local Institution - 780, Telavi
- Germany (19):
  - Local Institution - 629, Berlin
  - Local Institution - 653, Berlin
  - Local Institution - 648, Berlin
  - Local Institution - 628, Berlin
  - Local Institution - 664, Brandenburg
  - Local Institution - 732, Dachau
  - Local Institution - 574, Frankfurt am Main
  - Local Institution - 657, Frankfurt am Main
  - Local Institution - 658, Halle
  - Local Institution - 656, Halle
  - Local Institution - 652, Hamburg
  - Local Institution - 591, Hanover
  - Local Institution - 649, Keil
  - Local Institution - 337, Leipzig
  - Local Institution - 660, Mainz
  - Local Institution - 667, Münster
  - Local Institution - 620, Neuruppin
  - Local Institution - 584, Nürtingen
  - Local Institution - 661, Stuttgart
- Greece (8):
  - Local Institution - 790, Athens
  - Local Institution - 588, Athens
  - Local Institution - 791, Athens
  - Local Institution - 792, Athens
  - Local Institution - 592, Athens, Attiki
  - Local Institution - 787, Heraklion
  - Local Institution - 789, Thessaloniki
  - Local Institution - 788, Thessaloniki
- Hong Kong (2):
  - Local Institution - 404, Hong Kong
  - Local Institution - 405, Kowloon
- Hungary (11):
  - Local Institution - 798, Békéscsaba
  - Local Institution - 803, Budapest
  - Local Institution - 804, Budapest
  - Local Institution - 556, Budapest
  - Local Institution - 801, Győr
  - Local Institution - 555, Gyula
  - Local Institution - 797, Miskolc
  - Local Institution - 800, Nagykanizsa
  - Local Institution - 816, Szekszárd
  - Local Institution - 805, Szentes
  - Local Institution - 799, Székesfehérvár
- Israel (7):
  - Local Institution - 343, Afula
  - Local Institution - 346, Beer Jacob
  - Local Institution - 350, Haifa
  - Local Institution - 347, Jerusalem
  - Local Institution - 349, Kfar Saba
  - Local Institution - 341, Petah Tikva
  - Local Institution - 340, Tel Aviv
- Lithuania (5):
  - Local Institution - 605, Kaunas
  - Local Institution - 603, Klaipėda
  - Local Institution - 607, Vilnius
  - Local Institution - 606, Vilnius
  - Local Institution - 604, Vilnius
- Netherlands (6):
  - Local Institution - 952, Amsterdam
  - Local Institution - 955, Amsterdam
  - Local Institution - 956, Groningen
  - Local Institution - 949, Nijmegen
  - Local Institution - 951, Sittard-Geleen
  - Local Institution - 954, Tilburg
- Poland (27):
  - Local Institution - 580, Częstochowa
  - Local Institution - 988, Elblag
  - Local Institution - 579, Gdansk
  - Local Institution - 978, Gdansk
  - Local Institution - 577, Gdynia
  - Local Institution - 906, Jelenia Góra
  - Local Institution - 757, Józefów
  - Local Institution - 578, Katowice
  - Local Institution - 834, Ksawerów
  - Local Institution - 581, Lodz
  - Local Institution - 981, Lodz
  - Local Institution - 976, Nowy Targ
  - Local Institution - 963, Rzeszów
  - Local Institution - 979, Sopot
  - Local Institution - 835, Szczecin
  - Local Institution - 586, Warsaw
  - Local Institution - 833, Warsaw
  - Local Institution - 989, Warsaw
  - Local Institution - 807, Warsaw
  - Local Institution - 893, Wierzchosławice
  - Local Institution - 983, Wroclaw
  - Local Institution - 984, Wroclaw
  - Local Institution - 582, Wroclaw
  - Local Institution - 982, Wroclaw
  - Local Institution - 831, Wroclaw
  - Local Institution - 987, Wroclaw
  - Local Institution - 832, Wroclaw
- Portugal (4):
  - Local Institution - 959, Coimbra
  - Local Institution - 958, Guimarães
  - Local Institution - 961, Loures
  - Local Institution - 957, Viana do Castelo
- Russia (34):
  - Local Institution - 966, Barnaul
  - Local Institution - 871, Barnaul
  - Local Institution - 589, Bataysk
  - Local Institution - 621, Chelyabinsk
  - Local Institution - 991, Chelyabinsk
  - Local Institution - 998, Kaliningrad
  - Local Institution - 882, Kaluga
  - Local Institution - 849, Kemerovo
  - Local Institution - 566, Moscow
  - Local Institution - 995, Moscow
  - Local Institution - 873, Moscow
  - Local Institution - 870, Moscow
  - Local Institution - 869, Moscow
  - Local Institution - 990, Nizhny Novgorod
  - Local Institution - 853, Novosibirsk
  - Local Institution - 876, Novosibirsk
  - Local Institution - 996, Omsk
  - Local Institution - 875, Orenburg
  - Local Institution - 867, Penza
  - Local Institution - 863, Saint Petersburg
  - Local Institution - 993, Saint Petersburg
  - Local Institution - 868, Saint Petersburg
  - Local Institution - 857, Saint Petersburg
  - Local Institution - 879, Saint Petersburg
  - Local Institution - 878, Saint Petersburg
  - Local Institution - 874, Saint Petersburg
  - Local Institution - 865, Samara
  - Local Institution - 992, Saratov
  - Local Institution - 866, Sochi
  - Local Institution - 877, Tomsk
  - Local Institution - 881, Ufa
  - Local Institution - 880, Volgograd
  - Local Institution - 583, Yekaterinburg
  - Local Institution - 872, Yekaterinburg
- Local Institution - 546, Cape Town, Senegal
- Serbia (9):
  - Local Institution - 887, Belgrade
  - Local Institution - 596, Belgrade
  - Local Institution - 886, Belgrade
  - Local Institution - 890, Belgrade
  - Local Institution - 891, Kragujevac
  - Local Institution - 884, Novi Sad
  - Local Institution - 885, Pančevo
  - Local Institution - 585, Vršac
  - Local Institution - 889, Zrenjanin
- Slovakia (7):
  - Local Institution - 900, Bratislava
  - Local Institution - 894, Bratislava
  - Local Institution - 895, Brezno
  - Local Institution - 899, Nitra
  - Local Institution - 897, Nové Zámky
  - Local Institution - 898, Prešov
  - Local Institution - 896, Rimavská Sobota
- Local Institution - 904, Celje, Slovenia
- South Africa (7):
  - Local Institution - 543, Gauteng
  - Local Institution - 545, Kempton Park
  - Local Institution - 544, Pretoria
  - Local Institution - 542, Pretoria
  - Local Institution - 549, Pretoria
  - Local Institution - 548, Somerset West
  - Local Institution - 547, Val de Grace
- South Korea (5):
  - Local Institution - 434, Busan
  - Local Institution - 431, Busan
  - Local Institution - 432, Daegu
  - Local Institution - 438, Seoul
  - Local Institution - 429, Suwon
- Spain (8):
  - Teknon Medical Center, Barcelona
  - University Hospital Reina Sofia, Córdoba
  - University Hospital of Girona Dr. Josep Trueta, Girona
  - Hospital Universitario De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Local Institution - 695, Madrid
  - University Hospital Puerta de Hierro Majadajonda, Majadahonda, Madrid
  - University Hospital Marques de Valdecilla (HUMV), Santander
  - Local Institution - 697, Valencia
- Local Institution - 625, Stockholm, Sweden
- Taiwan (7):
  - Local Institution - 460, Kaohsiung City
  - Local Institution - 463, Kaohsiung, San Ming Dist.
  - Local Institution - 461, Niao-Sung Hsiang Kaohsiung County
  - Local Institution - 459, Tainan, Taiana
  - Local Institution - 462, Taoyuan
  - Local Institution - 464, Tapei, Beitou Dist.
  - Local Institution - 465, Tapei
- Turkey (Türkiye) (5):
  - Local Institution - 357, Ankara
  - Local Institution - 365, Elâzığ
  - Local Institution - 358, Istanbul
  - Local Institution - 361, Istanbul
  - Local Institution - 353, Kadiköy/Istanbul
- Ukraine (16):
  - Local Institution - 922, Chernivtsi
  - Local Institution - 929, Ivano-Frankivsk
  - Local Institution - 965, Kharkiv
  - Local Institution - 920, Khmelnytskyi
  - Local Institution - 933, Kropyvnytskyi
  - Local Institution - 923, Kyiv
  - Local Institution - 563, Kyiv
  - Local Institution - 564, Kyiv
  - Local Institution - 977, Kyiv
  - Local Institution - 590, Lutsk
  - Local Institution - 974, Lviv
  - Local Institution - 902, Odesa
  - Local Institution - 932, Vinnytsia
  - Local Institution - 924, Vinnytsia
  - Local Institution - 587, Zaporizhia
  - Local Institution - 925, Zaporizhzhya

REFERENCES:
- [Derived] Feagan BG, Schreiber S, Afzali A, Rieder F, Hyams J, Kollengode K, Pearlman J, Son V, Marta C, Wolf DC, D'Haens GG. Ozanimod as a novel oral small molecule therapy for the treatment of Crohn's disease: The YELLOWSTONE clinical trial program. Contemp Clin Trials. 2022 Nov;122:106958. doi: 10.1016/j.cct.2022.106958. Epub 2022 Oct 5. PMID 36208720
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozanimod: Participants with moderate to severe acute Crohn's disease were administered Ozanimod capsule orally. Participants were administered 0.23 milligram (mg) of Ozanimod capsule (daily) from Day 1 to Day 4 followed by 0.46 mg of Ozanimod (2 capsules of 0.23 mg daily) from Day 5 to Day 7 followed by 0.92 mg of Ozanimod capsule (daily) from Day 8 to Week 12.
- Placebo: Participants with moderate to severely active Crohn's disease were orally administered Placebo (daily) from Day 1 to Week 12.
Period: Overall Study
Arm/Group | Ozanimod | Placebo
Started (Intent to Treat population includes all the randomized participants.) | 403 | 203
Safety Population (Subjects who received at least 1 dose of study drug.) | 404 (1 participant earlier randomized or pre-assigned to Placebo arm in error received Ozanimod) | 202
Completed | 360 | 183
Not Completed | 43 | 20
Not completed — Other Reason | 4 | 1
Not completed — Site Closed | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Lack of Efficacy | 9 | 2
Not completed — Adverse Event | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozanimod | Placebo | Total
Number analyzed (Participants) | 403 | 203 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.69) | 37.7 (13.79) | 39.1 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 90 | 272
  Male | 221 | 113 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 378 | 188 | 566
  Unknown or Not Reported | 12 | 3 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 329 | 166 | 495
  BLACK OR AFRICAN AMERICAN | 7 | 1 | 8
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 1
  ASIAN | 47 | 29 | 76
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 1
  OTHER | 8 | 4 | 12
  NOT REPORTED | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Score < 150
Description: The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Week 12
Population: Intent to Treat population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 29.8 | 30.5
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.8125, Cochran-Mantel-Haenszel; Odds ratio, and p-value are obtained using the CMH test stratified by corticosteroid use at baseline (yes or no), and prior biologic use (yes or no); Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.66 to 1.39]

2. Secondary Outcome: Percentage of Participants With Abdominal Pain and Stool Frequency Clinical Remission
Description: Abdominal pain and stool frequency clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤ 3 with abdominal pain and stool frequency no worse than baseline at Week 12. Participants entered the responses in diaries daily. The 7 days entries prior to Week 12 visit were considered for calculating average abdominal pain score and stool frequency. The abdominal pain was graded on severity of 0 (none) to 3 (severe) scale and stool frequency was defined number of liquid or soft stools per day. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Time Frame: Week 12
Population: Intent to Treat Population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 29.0 | 26.6
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.5400, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.77 to 1.66]

3. Secondary Outcome: Percentage of Participants With a Simple Endoscopic Score for Crohn's Disease (SES-CD) Score Decrease From Baseline of ≥ 50%
Description: The SES-CD assessed the degree of inflammation. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater degree of inflammation. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Time Frame: Week 12
Population: Intent to Treat population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 25.6 | 21.2
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.2411, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.85 to 1.95]

4. Secondary Outcome: Percentage of Participants With Reduction From Baseline in the Crohn's Disease Activity Index (CDAI) Score of >= 100 Points or a Total CDAI Score < 150
Description: The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease (CD). The CDAI uses a questionnaire with 8 disease activity variables: number of soft/liquid stools, severity of abdominal pain, general well-being, presence of complications, need for antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. The sub scores of number of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Time Frame: Week 12
Population: Intent to treat population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 46.2 | 47.3
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.7469, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.67 to 1.34]

5. Secondary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Score Reduction From Baseline of ≥ 100 Points or CDAI Score < 150 and SES-CD Decrease From Baseline of ≥ 50%
Description: CDAI include 8 components number of soft/liquid stools, severity of abdominal pain, wellbeing, complications, need antidiarrheal drugs, abdominal mass, hematocrit, deviation in body wt. Subscores of numbers of soft/liquid stool, severity of abdominal pain (0 [none] to 3 [Severe]), general well-being (0 [well] to 4 [terrible] were summed over the 7 days prior to visit. The others weighted to create the total CDAI score ranging 0-600 with higher score indicating worse outcome. The SES-CD has 4 components size of ulcers, ulcerated surface, affected surface, presence of narrowing. Each component was scored on scale of 0 (none) to 3 (worst). In SES-CD, each of 4 components are assessed in the five segments: ileum, right, transverse, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for overall, with larger scores show greater degree of inflammation.
Time Frame: Week 12
Population: Intent to Treat population included all the randomized participants. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 16.9 | 14.3
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.4255, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.75 to 1.97]

6. Secondary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Score < 150 and Simple Endoscopic Score for Crohn's Disease (SES-CD) Score Decrease From Baseline of ≥ 50%
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 11.7 | 11.3
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.9313, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.60 to 1.76]

7. Secondary Outcome: Percentage of Participants With Abdominal Pain and Stool Frequency Clinical Remission and a Simple Endoscopic Score for Crohn's Disease (SES-CD) Score <= 4 Points and Decrease >= 2 Points
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤ 3 times with AP and SF no worse than baseline at Week 12. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. The AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day. The SES-CD has 4 components size of ulcers, ulcerated surface, affected surface, presence of narrowing. Each component was scored on scale of 0 (none) to 3 (worst). In SES-CD, each of 4 components are assessed in the five segments: ileum, right, transverse, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for overall, with larger scores show greater degree of inflammation.
Time Frame: Week 12
Population: Intent to Treat population included all the randomized subjects. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 10.4 | 8.4
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.4339, Cochran-Mantel-Haenszel; Odds ratio and p-value are obtained using the CMH test stratified by corticosteroid use at baseline (yes or no), and prior biologic use (yes or no); Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.70 to 2.31]

8. Secondary Outcome: Percentage of Participants With Global Histologic Activity Score (GHAS) Remission
Description: GHAS assesses the inflammation and mucosal damage. GHAS has 8 components Epithelial damage, Architectural changes, Infiltration of mononuclear cells in the lamina propria, Infiltration of polymorphonuclear cells in the lamina propria, Polymorphonuclear cells in epithelium, Presence of erosion and/or ulcers, Presence of granuloma and number of biopsy specimens affected. Each of these components was scored on a scale of 0 (none/unaffected) to 2 (worst). Each of these 8 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. Within each segment, the GHAS score has a range of 0 - 16, and the total GHAS score has a range of 0 - 80. Higher numbers correspond to more inflammation and more mucosal damage. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Time Frame: Week 12
Population: Intent to treat population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 13.6 | 10.8
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.3330, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.77 to 2.20]

9. Secondary Outcome: Percentage of Participants With CDAI Reduction From Baseline of >=70 Points
Description: as for outcome 4
Time Frame: Week 12
Population: Intent to treat population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 52.9 | 51.7
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.8200, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.74 to 1.47]

10. Secondary Outcome: Percentage of Participants With Absence of Ulcers ≥ 0.5 cm With no Segment With Any Ulcerated Surface ≥10%
Description: The ulcerated surface were assessed via endoscopy.
Time Frame: Week 12
Population: Intent to treat participants included all the randomized participants.
Measure: Number; unit: percentage of partiicpants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of partiicpants | 25.3 | 24.1
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.7776, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.71 to 1.59]

11. Secondary Outcome: Percentage of Participants With a Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of ≥ 50%
Description: CDEIS is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon. The CDEIS divides the intestine into 5 segments: rectum, sigmoid and left colon, transverse colon, right colon, and ileum. Four variables are assessed in each segment: the presence of deep ulceration, the presence of superficial ulceration, the percentage of ulcerated surface, and the percentage of surface affected by CD, indicated on 10-cm visual analogue scales. In addition, the presence of ulcerated stenosis and the presence of nonulcerated stenosis are also assessed over the entire intestine. These factors are weighted and summed to calculate the total score ranging from 0- 44, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: Intent to Treat included all the randomized participants. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 27.5 | 21.7
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.1187, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.92 to 2.11]

12. Secondary Outcome: Percentage of Participants With Abdominal Pain (AP) and Stool Frequency (SF) Clinical Remission and an Endoscopic (50%) Response
Description: AP and SF clinical remission is average daily abdominal pain score ≤ 1 point, and average daily stool frequency ≤ 3 times with AP and SF no worse than baseline at Week 12. Participants entered responses in diaries daily. The 7 days entries prior to visit were considered for calculating average AP score and SF. AP was graded on severity of 0 (none) to 3 (severe) scale and SF was defined number of liquid or soft stools per day. SES-CD has 4 components size of ulcers, ulcerated surface, affected surface, presence of narrowing. Each component was scored on scale of 0 (none) to 3 (worst). Endoscopic Response is defined as >= 50% decrease from baseline in SES-CD. In SES-CD, each of 4 components are assessed in five segments: ileum, right, transverse, left colon, and rectum. The SES-CD was sum of individual scores of each of components across five segments. Range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for overall, with larger scores show greater degree of inflammation.
Time Frame: Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of particpants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of particpants | 11.7 | 9.4
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.4030, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.72 to 2.26]

13. Secondary Outcome: Percentage of Participants With Robarts Histologic Index (RHI) Mucosal Healing at Week 12
Description: RHI mucosal healing was defined as RHI remission combined with SES-CD <= 4 points and a SES-CD decrease from baseline >= 2 points with no SES-CD sub-score >1 point. RHI Remission is defined as no active inflammation in any measured segment. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 (none/unaffected) to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater degree of inflammation.
Time Frame: Week 12
Population: Intent-to-treat population included all the randomized participants. Baseline was defined as the last assessment prior to the start time of the first drug administration if time of measurement is available else the last assessment prior to or on the date of the first drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Ozanimod | Placebo
Number analyzed (Participants) | 403 | 203
percentage of participants | 4.0 | 4.9
Statistical Analysis 1: Comparison: Ozanimod vs Placebo; Test type: Superiority; p = 0.5630, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.35 to 1.78]

ADVERSE EVENTS:
Time Frame: All cause mortality, non serious adverse events and serious adverse events were collected from the first dose and up to approximately 31 weeks.
Description: Treated population include all the participants who were treated with at least one dose of study drug. 1 participant earlier randomized or pre-assigned to Placebo arm in error received Ozanimod and was included in Ozanimod' arm.
Arm/Group | Ozanimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/404 | 0/202
Serious Adverse Events (participants affected / at risk) | 24/404 | 11/202
Other Adverse Events (participants affected / at risk) | 15/404 | 11/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod (N=404) | Placebo (N=202)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 10 | 6
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod (N=404) | Placebo (N=202)
Crohn's disease (Gastrointestinal disorders) | 15 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03440385/Prot_SAP_000.pdf